CLINICAL TRIAL: NCT02312050
Title: A Phase 2b, Placebo-Controlled, Randomized, Double-Blind, Multi-Center Study of GCS-100 in Patients With Chronic Kidney Disease Caused by Diabetes
Brief Title: A Phase 2b Study of GCS-100 in Patients With Chronic Kidney Disease Caused by Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LJ100-CKD04
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Chronic Kidney Disease
MeSH Terms: interventions — GCS-100

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GCS-100 1 mg (Experimental): Dose level 1 - administered via IV push injection weekly for 2 months, then every other week for an additional 4 months
  Interventions: Drug: GCS-100
- GCS-100 3 mg (Experimental): Dose level 2 - administered via IV push injection weekly for 2 months, then every other week for an additional 4 months
  Interventions: Drug: GCS-100
- GCS-100 9 mg (Experimental): Dose level 3 - administered via IV push injection weekly for 2 months, then every other week for an additional 4 months
  Interventions: Drug: GCS-100
- Normal Saline Solution 0.9% (Placebo Comparator): Placebo - administered via IV push injection weekly for 2 months, then every other week for an additional 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GCS-100 — 1 mg, 3 mg, or 9 mg IV push injections
  Arms: GCS-100 1 mg; GCS-100 3 mg; GCS-100 9 mg
Drug: Placebo
  Arms: Normal Saline Solution 0.9%

SUMMARY:
A phase 2b, placebo-controlled, randomized, double-blind, multi-center study of GCS-100 in patients with chronic kidney disease caused by diabetes. The study will enroll approximately 375 patients at multiple centers located in the United States. Study duration is 6 months. Patients will be randomly assigned 1:1:1:1 to treatment with placebo (0.9% Sodium Chloride Injection, USP), 1 mg, 3 mg, or 9 mg GCS-100. All doses of study drug will be administered via intravenous (IV) push injection once weekly for 2 months (8 weeks), then every other week for an additional 4 months (16 weeks).

DETAILED DESCRIPTION:
Galectin-3 contributes to fibrosis, is elevated in patients with ESRD, and correlates with adverse outcomes (de Boer et. al., 2011, Dang et. al., 2012, Fernandes Bertocchi et. al., 2008, Henderson et. al., 2008). Animal models with genetic knockout of galectin-3 demonstrate a reduction in structural and functional deficits in the kidney (Dang et. al., 2012, Fernandes Bertocchi et. al., 2008, Henderson et. al., 2008). GCS-100 is a galectin- 3 antagonist that has been shown to reduce fibrosis pre-clinically. Based on the role of galectin-3 and fibrosis in kidney disease, the Sponsor believes GCS-100 may be effective at treating patients with CKD caused by diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is capable of understanding the purpose and risks of the study and is able to provide written informed consent.
2. Patient is ≥ 18 and ≤ 90 years of age.
3. Patient has a baseline eGFR of 15 to < 45 mL/min/1.73m2, defined as the average of 2 measurements collected at Screening Visits 1 and 2, and determined using the 4-variable Modification of Diet in Renal Disease (MDRD) equation.
4. Patients with diabetic CKD diagnosis > 12 months, and if requiring renin-angiotensin-aldosterone system (RAAS) blockade medications, must be receiving stable doses (i.e., not requiring modification) for the 3 months prior to first study drug dose.
5. Stable eGFR as measured by a less than 25% variability of each Screening value from the average of the 2 Screening values taken no less than 5 days and no more than 10 days apart.
6. Patient is willing and able to comply with all protocol requirements.
7. Female patients of childbearing potential (i.e., women who have not been surgically sterilized or who have not been post-menopausal for at least 1 year) and male patients with partners of childbearing potential must agree to use medically acceptable methods of contraception throughout the study period.

Exclusion Criteria:

1. Treatment with an experimental (unlicensed) drug within 4 weeks prior to Screening visit 1.
2. Patients who are known to be allergic to citrus or have a history of any allergies associated with hypersensitivity to citrus.
3. Patients who have begun new treatment with angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), mineralocorticoid receptor blockers (MRBs), or direct renin inhibitors (DRIs) within the 3 months prior to first dose.
4. Kidney disease known to be due to causes other than diabetes.
5. Patients diagnosed with acute kidney injury (AKI) within the 3 months prior to first dose.
6. Planned renal replacement therapy of any kind within 6 months of first study drug dose.
7. Previous solid organ transplant.
8. Evidence of persistent, uncontrolled hypertension, i.e., systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg; or evidence of persistent, uncontrolled hypotension, i.e., systolic blood pressure ≤ 90 mmHg and diastolic blood pressure ≤ 40 mmHg at repeated measures during Screening.
9. Patients who have Screening clinical laboratory values of:

   1. Hemoglobin: ≤ 9 g/dL
   2. Total bilirubin: > 1.5X the upper limit of normal (ULN)
   3. ALT and/or AST: > 2.5X ULN
   4. HbA1c > 10.5%
10. Concomitant treatment with immunosuppressive agents, except for stable use of topical agents or inhaled steroids.
11. Patients who have previously received GCS-100 as part of another clinical trial.
12. Known history of cancer (excluding non-melanoma skin cancer that is not being actively treated) within 5 years of Screening.
13. Known history of human immunodeficiency virus, active hepatitis C virus (HCV), active hepatitis B virus (HBV), or prior history of infection with HBV (HBcAb positive); if adequate hepatic function has been documented for patients with HCV or prior history of hepatitis B without evidence of cirrhosis, the Medical Monitor may approve their enrollment.
14. Clinically relevant active infection and/or a serious co-morbid medical condition, such as recent myocardial infarction (within the last 6 months), unstable angina, difficult-to-control congestive heart failure, uncontrolled hypertension, difficult-to-control cardiac arrhythmias, severe or uncontrolled chronic obstructive or chronic restrictive pulmonary disease, and/or cirrhosis.
15. Patient had major surgery within 12 weeks of first study drug dose.
16. If female, patient is pregnant or breastfeeding.
17. Patient has a concomitant disease or condition, including laboratory abnormalities, which, in the opinion of the investigator, could interfere with the conduct of the study or put the patient at unacceptable risk.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The change in eGFR from Screening to measurements taken at Week 26 | 26 weeks

SECONDARY OUTCOMES:
Change in eGFR (as a scored value using 20% cut point) from Screening to Week 26 | 26 weeks
Change in eGFR (as a scored value using 30% cut point) from Screening to Week 26 | 26 weeks
Incidence of renal replacement therapy (RRT) | 26 weeks
Incidence of major cardiac events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George F Tidmarsh, MD, PhD, Study Director — La Jolla Pharmaceutical Company
Locations (8):
- United States (8):
  - Balboa Nephrology Medical Group, Chula Vista, California
  - Balboa Nephrology Medical Group, El Centro, California
  - Balboa Nephrology Medical Group, La Jolla, California
  - California Institute for Renal Research, La Mesa, California
  - Denver Nephrology, Denver, Colorado
  - Mountain Kidney & Hypertension, Asheville, North Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Clinical Advancement Center, San Antonio, Texas